CLINICAL TRIAL: NCT03970252
Title: A Pilot and Feasibility Study of PD-1 Blockade With Nivolumab in Combination With Chemotherapy in Patients With Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: Nivolumab in Combination With Chemotherapy Pre-Surgery in Treating Patients With Borderline Resectable Pancreatic Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-000290; NCI-2019-02886 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma; Resectable Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; Nivolumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (nivolumab, mFOLFIRINOX) (Experimental): Patients receive nivolumab IV over 60 minutes on day 1. Patients also receive fluorouracil IV over 10 minutes and over 46 hours, irinotecan hydrochloride IV over 90-120 minutes, leucovorin calcium IV over 120 minutes, and oxaliplatin IV over 120 minutes on days 1 and 15. Treatments repeat every 28 days for 3-6 cycles in the absence of disease progression or unacceptable toxicity. Within 2-4 weeks after treatment, patients with resectable disease undergo surgery. Within 8-12 weeks after surgery, patients with successful resection may receive 6 additional cycles of fluorouracil, irinotecan hydrochloride, leucovorin calcium, and oxaliplatin in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan; Drug: Irinotecan Hydrochloride; Drug: Leucovorin; Drug: Leucovorin Calcium; Biological: Nivolumab; Drug: Oxaliplatin; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Irinotecan — Given IV
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This pilot and feasibility study studies how well nivolumab and combination chemotherapy work before surgery in treating patients with pancreatic cancer that could possibly be removed by surgery. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body?s immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as fluorouracil, irinotecan hydrochloride, leucovorin calcium and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab in combination with chemotherapy before surgery may work better in treating patients with pancreatic cancer compared to chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate development of clinically relevant pancreatic fistula in the post-operative period after neoadjuvant treatment with nivolumab and fluorouracil, irinotecan hydrochloride, leucovorin calcium and oxaliplatin (FOLFIRINOX) (FFX).

II. To evaluate pathologic complete response after neoadjuvant nivolumab and FOLFIRINOX (FFX).

SECONDARY OBJECTIVES:

I. To evaluate early efficacy measured by percent change of CA 19-9 response rate, R0 resection rate, overall response rate (ORR) and disease free survival (DFS).

EXPLORATORY OBJECTIVES, OTHER ASSESSMENTS:

I. To determine degree of changes in the tumor microenvironment (TME) of nivolumab and modified (m) FFX on cell proliferation and apoptosis.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 60 minutes on day 1. Patients also receive fluorouracil IV over 10 minutes and over 46 hours, irinotecan hydrochloride IV over 90-120 minutes, leucovorin calcium IV over 120 minutes, and oxaliplatin IV over 120 minutes on days 1 and 15. Treatments repeat every 28 days for 3-6 cycles in the absence of disease progression or unacceptable toxicity. Within 2-4 weeks after treatment, patients with resectable disease undergo surgery. Within 8-12 weeks after surgery, patients with successful resection may receive 6 additional cycles of fluorouracil, irinotecan hydrochloride, leucovorin calcium, and oxaliplatin in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic adenocarcinoma
* One of the following:

  * Borderline resectable disease. There are multiple definitions of borderline resectable pancreatic ductal adenocarcinoma (PDAC) including the MD Anderson definition and the criteria developed during the Consensus Conference sponsored by the American Hepato-Pancreato-Biliary Association, Society of Surgical Oncology, and Society for Surgery of the Alimentary Tract. Borderline resectable PDAC cases will be identified per the definition developed in the currently running inter-group pilot trial for borderline resectable pancreatic cancer (NCT01821612). Per this trial, borderline resectable PDAC is defined as the presence of any one or more of the following on computed tomography (CT):

    * An interface between the primary tumor and the superior mesenteric vein or portal vein (SMV-PV) measuring >= 180 degrees of the circumference of the vessel wall
  * Short-segment occlusion of the SMV-PV with normal vein above and below the level of obstruction that is amenable to resection and venous reconstruction
  * Short segment interface (of any degree) between tumor and hepatic artery with normal artery proximal and distal to the interface that is amenable to resection and reconstruction
  * An interface between the tumor and superior mesenteric artery (SMA) measuring < 180 degrees of the circumference of the vessel wall
* Performance status of Eastern Cooperative Oncology Group (ECOG) of 0-1
* Therapy naive
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dl
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) and aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Serum creatinine (sCr) =< 1.5 x ULN or creatinine clearance (Ccr) >= 40 mL/min as calculated by the modified Cockcroft-Gault formula
* Peripheral neuropathy < grade 2

Exclusion Criteria:

* Locally advanced (clearly unresectable) or metastatic disease
* Known status of human immunodeficiency virus (HIV) which is not well-controlled at the time of study eligibility
* Untreated hepatitis B infection
* Active infection or antibiotics within 48 hours prior to study
* Currently active second primary malignancy or history of malignancy less than 5 years prior to the time of study eligibility (patients with history of skin cancers excluding melanoma will be eligible for participation)
* Serious medical comorbidities such as New York Heart Association class III/IV cardiac disease, uncontrolled cardiac arrhythmias, myocardial infarction over the past 12 months
* Known, existing uncontrolled coagulopathy. Patients who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation are eligible IF: they are appropriately anticoagulated and have not had a grade 2 or greater bleeding episode in the 3 weeks before day 1
* Prior history of cerebrovascular accident or transient ischemic attack, or pre-existing carotid artery disease
* Known pregnancy, nursing women or positive pregnancy test. Requirement for women of childbearing potential (WOCBP) must have a pregnancy test every 4 weeks and WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab
* Any prisoners, or subjects who are compulsory detained are excluded
* Any condition that would preclude informed consent, consistent follow-up and compliance for the study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Clinically relevant pancreatic fistula in the post-operative period after neoadjuvant treatment with nivolumab and fluorouracil, irinotecan hydrochloride, leucovorin calcium and oxaliplatin (FOLFIRINOX) (mFFX) chemotherapy | Up to 3 years
  Descriptive statistics with frequency and proportion will be used.
Pathologic complete response after nivolumab and mFFX treatment | Up to 3 years
  Descriptive statistics with frequency and proportion will be used.

SECONDARY OUTCOMES:
Percent change of CA 19-9 response rate | Baseline up to 3 years
  Descriptive statistics with frequency and proportion will be used to analyze the CA19-9 response rate.
R0 resection rate | Up to 3 years
Overall response rate (ORR) | Up to 3 years
  Descriptive statistics with frequency and proportion will be used to analyze ORR.
Disease free survival (DFS) | Up to 3 years
  Kaplan-Meier methods will be used to analyze DFS with median and 95% confidence interval (CI).
Incidence of adverse events | Up to 28 days after last dose of study drug
  Will be categorized and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.3.
Delayed wound healing | Up to 3 years
Wound dehiscence | Up to 3 years
Wound infection | Up to 3 years

OTHER OUTCOMES:
Changes in immune cell infiltrates and cancer cell IFNgamma signaling in response to FOLFIRINOX and nivolumab treatment | Baseline up to 3 years
  Will examine the tissue from baseline to post-therapy at the time of surgery or at the time of progression. Will use descriptive statistics and graphical displays to compare the percent change in stromal depletion overall and to describe the association with cell proliferation and death. In addition, will graphically explore the percent change in stromal depletion for patients who undergo surgery compared to those who have disease progression.
Signaling and metabolomic changes in pancreatic ductal adenocarcinoma (PDAC) cancer cells that respond to IFNgamma | Baseline up to 3 years
  Will examine the tissue from baseline to post-therapy at the time of surgery or at the time of progression. Will use descriptive statistics and graphical displays to compare the percent change in stromal depletion overall and to describe the association with cell proliferation and death. In addition, will graphically explore the percent change in stromal depletion for patients who undergo surgery compared to those who have disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Zev A Wainberg, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States